CLINICAL TRIAL: NCT02193009
Title: SipSmarter: A Nutrition Literacy Approach to Reducing Sugary Beverages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: University of Kansas (Other); University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA154364 (NIH)
Record Dates: First submitted 2014-07-11; First posted 2014-07-17 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Dietary Habits; Physical Activity
MeSH Terms: conditions — Feeding Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIPsmartER, behavioral intervention (Experimental): Aimed at decreasing sugar-sweetened beverage consumption
  Interventions: Behavioral: SipSmarter
- Move More, behavioral intervention (Active Comparator): Aimed at physical activity promotion
  Interventions: Behavioral: MoveMore

INTERVENTIONS:
Behavioral: SipSmarter — 6-month behavioral trial
  Arms: SIPsmartER, behavioral intervention
Behavioral: MoveMore — 6 month behavioral trial
  Arms: Move More, behavioral intervention

SUMMARY:
The primary aim of this pragmatic randomized-controlled trial was to determine the effectiveness of a scalable 6-month intervention aimed at decreasing SSB consumption (SIPsmartER) when compared to a matched contact physical activity promotion control group (MoveMore).

DETAILED DESCRIPTION:
The primary aim of this application targeting at-risk residents from rural southwest Virginia counties is to:

1. Determine the effectiveness of SIPsmart and SIPsmartER at decreasing SSB consumption when compared to a matched contact control group targeting walking behaviors.

The secondary aims are to:

1. Explore causal pathways through which changes in SSB attitudes, subjective norms, and perceived behavioral control influence behavioral intentions and SSB consumption, and the extent to which changes in SSB consumption are mediated by changes in nutrition numeracy and nutrition-related media literacy.
2. Determine the reach and representativeness, adoption feasibility, degree to which the intervention was implemented as intended (and associated costs), and the maintenance of behavior changes 6 and 12 months post intervention (i.e., 18 months from baseline) when compared to control.
3. Assess intervention impacts on body weight.

An exploratory aim is to:

1. Assess intervention impacts on a 13C biomarker, a new non-invasive biomarker fingerstick technique for added sugar intake, and evaluate the changes in this biomarker over time.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included English-speaking adults >18 years of age, who consume >200 SSB kcals/day, self-report no contraindications for physical activity, and have regular access to a telephone.

Exclusion Criteria:

* To minimize potential confounds, only one member per household is eligible to enroll and individuals cannot be concurrently enrolled in a Cooperative Extension program because these programs focus on improving nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2011-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Kilocalories of Sugar-Sweetened Beverages at 6 months | baseline, 6-months

SECONDARY OUTCOMES:
Change from Baseline in Minutes of Physical Activity at 6 months | baseline, 6-months

OTHER OUTCOMES:
Change from Baseline in Weight at 6 months | baseline, 6-months
Change from Baseline in C13 biomarker at 6 months | baseline, 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Zoellner, PhD, RD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Departmen of Human Nutrition, Foods, and Exercise, Blacksburg, Virginia, United States

REFERENCES:
- [Derived] Zoellner JM, You W, Estabrooks PA, Chen Y, Davy BM, Porter KJ, Hedrick VE, Bailey A, Kruzliakova N. Supporting maintenance of sugar-sweetened beverage reduction using automated versus live telephone support: findings from a randomized control trial. Int J Behav Nutr Phys Act. 2018 Oct 4;15(1):97. doi: 10.1186/s12966-018-0728-7. PMID 30286755
- [Derived] Kruzliakova N, Estabrooks PA, You W, Hedrick V, Porter K, Kiernan M, Zoellner J. The Relationship Between the Stanford Leisure-Time Activity Categorical Item and the Godin Leisure-Time Exercise Questionnaire Among Rural Intervention Participants of Varying Health Literacy Status. J Phys Act Health. 2018 Apr 1;15(4):269-278. doi: 10.1123/jpah.2017-0284. Epub 2018 Feb 9. PMID 29421974
- [Derived] Hedrick VE, Davy BM, You W, Porter KJ, Estabrooks PA, Zoellner JM. Dietary quality changes in response to a sugar-sweetened beverage-reduction intervention: results from the Talking Health randomized controlled clinical trial. Am J Clin Nutr. 2017 Apr;105(4):824-833. doi: 10.3945/ajcn.116.144543. Epub 2017 Mar 1. PMID 28251935
- [Derived] Estabrooks P, You W, Hedrick V, Reinholt M, Dohm E, Zoellner J. A pragmatic examination of active and passive recruitment methods to improve the reach of community lifestyle programs: The Talking Health Trial. Int J Behav Nutr Phys Act. 2017 Jan 19;14(1):7. doi: 10.1186/s12966-017-0462-6. PMID 28103935
- [Derived] Zoellner JM, Hedrick VE, You W, Chen Y, Davy BM, Porter KJ, Bailey A, Lane H, Alexander R, Estabrooks PA. Effects of a behavioral and health literacy intervention to reduce sugar-sweetened beverages: a randomized-controlled trial. Int J Behav Nutr Phys Act. 2016 Mar 22;13:38. doi: 10.1186/s12966-016-0362-1. PMID 27000402
- [Derived] Hedrick VE, Zoellner JM, Jahren AH, Woodford NA, Bostic JN, Davy BM. A Dual-Carbon-and-Nitrogen Stable Isotope Ratio Model Is Not Superior to a Single-Carbon Stable Isotope Ratio Model for Predicting Added Sugar Intake in Southwest Virginian Adults. J Nutr. 2015 Jun;145(6):1362-9. doi: 10.3945/jn.115.211011. Epub 2015 Apr 8. PMID 25855120